CLINICAL TRIAL: NCT00340834
Title: A 12-month Double-blind, Randomized, Multicenter, Active-controlled, Parallel-group Study Comparing the Efficacy and Safety of 0.5 mg and 1.25 mg Fingolimod (FTY720) Administered Orally Once Daily Versus Interferon ß-1a (Avonex) Administered im Once Weekly in Patients With Relapsing-remitting Multiple Sclerosis With Optional Extension Phase
Brief Title: Efficacy and Safety of Fingolimod in Patients With Relapsing-remitting Multiple Sclerosis With Optional Extension Phase
Acronym: TRANSFORMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2302; CFTY720D2302E1 (Other: Novartis)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: FTY720; Interferon; RRMS; Multiple Sclerosis; Efficacy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- Fingolimod 1.25 mg (Experimental)
  Interventions: Drug: Fingolimod 1.25 mg
- Fingolimod 0.5 mg (Experimental)
  Interventions: Drug: Fingolimod 0.5 mg
- Interferon β-1a 30 µg (Active Comparator)
  Interventions: Drug: Interferon β-1a 30 µg

INTERVENTIONS:
Drug: Fingolimod 1.25 mg — Core: Patients self-administered fingolimod 1.25 mg capsules orally once daily. In addition, they self-administered an interferon β-1a placebo intramuscular (im) injection once weekly.
  Extension: Patients self-administered fingolimod 1.25 mg capsules orally once daily until switched to 0.5 mg capsules upon study protocol amendment.
  Other Names: FTY720
  Arms: Fingolimod 1.25 mg
Drug: Fingolimod 0.5 mg — Core: Patients self-administered fingolimod 0.5 mg capsules orally once daily. In addition, they self-administered an interferon β-1a placebo intramuscular (im) injection once weekly.
  Extension: Patients self-administered fingolimod 0.5 mg capsules orally once daily.
  Other Names: FTY720
  Arms: Fingolimod 0.5 mg
Drug: Interferon β-1a 30 µg — Core: Patients self-administered interferon β-1a 30 μg in an intramuscular (im) injection once weekly. In addition, they self-administered a fingolimod placebo capsule orally once daily.
  Extension: Patients self-administered either fingolimod 1.25 mg or 0.5 mg capsules orally once daily until switched to 0.5 mg capsules upon study protocol amendment.
  Arms: Interferon β-1a 30 µg

SUMMARY:
This study assessed the safety, tolerability, and efficacy of 2 doses of oral fingolimod versus interferon β-1a to reduce the frequency of relapses in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages 18-55 with a diagnosis of multiple sclerosis (MS)
* Patients with a relapsing-remitting disease course
* Patients with Expanded Disability Status Scale (EDSS) score of 0-5.5

Exclusion Criteria:

* Patients with other chronic disease of the immune system, malignancies, acute pulmonary disease, cardiac failure, etc
* Pregnant or nursing women
* Patients who cannot tolerate treatment with an interferon

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1292 (Actual)
Dates: Start 2006-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmacuticals
Locations (167):
- United States (35):
  - North Central Neurology Associates, PC, 1809 Kress Street, Cullman, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - The Neurology Center, 3907 Waring Road, Suite 3, Oceanside, California
  - Associated Neurologists, PC, 69 Sand Pit Road, Suite 300, Danbury, Connecticut
  - Associated Neurologists of Southern CT, PC, 75 Kings Highway Cutoff, Fairfield, Connecticut
  - Yale University Multiple Sclerosis Center, New Haven, Connecticut
  - University of Florida Health Science Center, Jacksonville, Florida
  - Neurology Associates, PA, 301 N. Maitland Avenue, Suite A1, Maitland, Florida
  - University of Miami, Department of Neurology, Miami, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Roskamp Institute, 2040 Whitfield Ave., Sarasota, Florida
  - AMO Corporation, Tallahassee, Florida
  - Axiom Clinical Research of Florida, 2919 Swann Avenue, Suite 401, Tampa, Florida
  - University of South Florida, Department of Neurology, Tampa, Florida
  - The MS Center of Vero Beach, Vero Beach, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mid America Neuroscience Institute, 8550 Marshall Drive, Suite 100, Lenexa, Kansas
  - University Physician Group, #1 Barnes-Jewish Hospital Plaza, Suite 16304, St Louis, Missouri
  - Neuroscience and Spine Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, 1540 Sunday Drive, Raleigh, North Carolina
  - Neurology & Neuroscience Associates, Inc, Akron, Ohio
  - Northern Ohio Neuroscience, LLC, Bellevue, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Neurology, Tualatin, Oregon
  - University of Pittsburgh, Department of Neurology, Pittsburgh, Pennsylvania
  - Absher Neurology, 274-A Commonwealth Drive, Greenville, South Carolina
  - Mountain Empire Neurological Associates, PC, 3183 West State Street, Suite 1201, Bristol, Tennessee
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Private Practice, 3815 23rd Street, Lubbock, Texas
  - Integra Clinical Research, 4242 Medical Drive, Suite 6100, San Antonio, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
  - Rockwood Clinic, P.S., Spokane, Washington
  - West Virginia University Health Associates, Morgantown, West Virginia
  - Center for Neurological Disorders - Aurora St. Luke's Med Center, Milwaukee, Wisconsin
- Argentina (7):
  - Ineba, Guarda Vieja 4435, Capital Federal, Buenos Aires
  - Fundacion Rosarina de Neurorehabilitacion, Rosario, Santa Fe Province
  - Instituto de Neurociencias de Rosario, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundacion Lenox Cordoba, Córdoba
  - Hospital J. M. Ramos Mejia, General Urquiza 609, Buenos Aires
  - FLENI, Montaneses 2325, Buenos Aires
- Australia (7):
  - Strategic Health Evaluators, Chatswood, New South Wales
  - Royal Prince Alfred Hospital, Department of Medicine, Level, Missenden R, Camperdown, New South Wales
  - Liverpool Hospital, Neurology Department, Health Services Building, 4th Floor, Goulburn and Campbell Street, Liverpool, New South Wales
  - Gosford Private Hospital, North Gosford, New South Wales
  - St George Private Hospital, Suite 7E, Level 5, South Street, Kogarah, New South Wales
  - Box Hill Hopsital, Level 3, 16 Arnold Street, Box Hill, Victoria
  - Royal Melbourne Hospital, Suite 30, Grattan St., Parkbville, Victoria
- Austria (6):
  - Landesklinikum St. Poelten, Probst-Ruehrer-Str. 4, Sankt Pölten, Sankt Poelten
  - Landes-Narvenklinik Wagner-Jauregg, Abteilung Fuer Neurologie, Linz
  - Universitätsklinik f. Neurologie Innsbruck, Anichstrasse 35, Innsbruck
  - Landes-Nervenklinik Christian Doppler Klinik, Ignaz Harrerstr. 79 , Salzburg
  - Evangel.Krankenh./Wien-Waehring Außenstelle, Vienna
  - Univ.-Klinik fuer Neurologie AKH, Vienna
- Belgium (4):
  - Cliniques Universitaires Saint Luc, Avenue Hippocrate 10, Bruxelles
  - UZ Brussel, Laarbeeklaan 101, Brussels
  - Nationaal Multiple Sclerose Centrum v.z.w, Melsbroek
  - Regionaal Ziekenhuis Sint-Trudo - Campus Sint-Jozef, Sint-Truiden
- Brazil (6):
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Hospital das Clincas - UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas da FMRPUSP, Ribeirão Preto, São Paulo
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital dos Servidores do Estado, Rio de Janeiro
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro
- Canada (9):
  - Fraser Health MS Clinic, Burnaby Hospital, 3935 Kincaid Street, Vancouver, British Columbia
  - UBC MS Research, 2211 Westbrook Mall, Vancouver, British Columbia
  - Nepean Medical Centre, 1 Centrepointe Drive, Suite 407, Ottawa, Ontario
  - St. Michael's Hospital, Chief, Division of Neurology, 30 Bond Street,Suite 3007 - Shuter Wing, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, 3001 12th Avenue North, Fleurimont, Quebec
  - Charles Lemoyne Hospital, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Montreal Neurological Institute, 3801 University Street, Montreal, Quebec
  - The Ottawa General Hospital, 501 Smyth Rd., Ottawa
- Egypt (5):
  - Private Clinic, 48 Sidi Gaber St., Alexandria
  - 35, Dokki St., Apt. 4, Cairo
  - Al Azhar University, 11 Talaat Harb St, Fourth Floor, Apt 18, Cairo
  - Private Clinic, 35 Dokki St., Apt. 4, Cairo
  - Private Clinic, 7 Batal Ahmed Abdelaziz St Abdeen, Cairo
- France (6):
  - Hopital La Timone Cpcet, Rue Jean Moulin, Marseille
  - Hopital Central, 29 Avenue du Marechal de Lattre de Tassigny, Nancy
  - Hôpital Pellegrin, Place Amélie Raba Léon, Bordeaux Cedex
  - Hopital De Purpan, Place Du Dr. Baylac, Toulouse Cedex
  - Centre Hospitalier de Poissy, 10 rue du Champ Gaillard, Poissy
  - Hoppital Pasteur, Archet II, 30 avenue de la Voie, Romaine
- Germany (25):
  - Investigational Site, Bamberg
  - Investigational Site, Berlin
  - Investigational Site, Bremen
  - Investigational Site, Buchholz
  - Investigational Site, Cologne
  - Investigational Site, Dresden
  - Investigational Site, Düsseldorf
  - Investigational Site, Erbach/Odenwald
  - Investigational Site, Essen
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Greifswald
  - Investigational Site, Hamburg
  - Investigational Site, Hanover
  - Investigational Site, Heidelberg
  - Investigational Site, Hennigsdorf
  - Investigational Site, Lengerich
  - Investigational Site, Mainz
  - Investigational Site, München
  - Investigational Site, Potsdam
  - Investigational Site, Teupitz
  - Investigational Site, Trier
  - Investigational Site, Tübingen
  - Investigational Site, Ulm
  - Investigational Site, Wermsdorf
  - Investigational Site, Würzburg
- Greece (6):
  - Univ. Hospital of Heraklion, Voutes, Heraklion, Crete
  - Errikos Dinan General Hospital, 107 Mesogion Ave., Athens
  - General Hospital of Athens G. Gennimatas, 154 Mesogeion Ave., Athens
  - Metropolitan Hospital, Ethnarchou Makariou 6 & Eleftheriou Venizelou 1, Athens
  - General University Hospital of Patra-RIO, Patra - RIO
  - Ahepa University General Hospital of Thessaloniki, 1 Stilp. Kyriakidi Str., Thessaloniki
- Hungary (6):
  - Debreceni Egyetem Orvos es Egszstd. Centr., Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Veszprem Megyei Csolnoky Ferenc Korhaz, Korhaz U. 1, Veszprem
  - Pecsi Tudomanyegyetem Neurologiai Klinika, Pécs
  - Peterfy Sandor u. Hospital, Neurology, U. 8-20m, Budapest
  - Uzsoki korhaz, Uzsoki U. 29., Budapest
- Italy (22):
  - Azienda Sanitaria Osp. S. Luigi, Gonzaga, Orbassano
  - Ospedale S. Antonio Abate, Via Pastori, 4, Gallarate, VA
  - Presidio Ospedaliero Roberto Binaghi, Cagliari
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Ferrara
  - Presidio Ospedaliero di Vaio Fidenza, Fidenza
  - Osp. Magg. Pol. Mangiagalli e Regina Elena - Fond. IRCCS, Milan
  - Az. Osp. Niguarda Ca' Granda, Milan
  - Presidio Ospedaliero di Montichiari, Montichiari
  - IRCCS Neurologico C. Mondino, Pavia
  - Az. Osp. Ospedale Consorziale e Policlinico, Piazza Giulio Cesare, 11 Bari
  - Az. Osp. Ospedale S. Martino - Università degli Studi, Via Antonio de Toni, 5, Genova
  - Ist. Neurol. Mediterraneo Neuromed, Via Atinense, 18, Pozzilli
  - Ospedali Riuniti Umberto I - GM Lancisi - G.Salesi, Via Conca, 71, Torrette Di Ancona
  - Osp. Clinicizzato Colle dell'Ara - Università G. D'Annunzio, Via Dei Vestini, 5 Chieti
  - Azienda Ospedaliera Sant'Andrea - Università La Sapienza, Via Di Grottarossa, 1035/1039, Roma
  - Azienda Ospedaliera di Padova - Università degli Studi, Via Giustiniani, 2, Padova
  - Az. Osp. Universitaria Policlinico Tor Vergata, Via Montpellier, 1, Roma
  - Ospedale San Raffaele - IRCCS, Via Olgettina, 48/60, Milano
  - Policlinico - Università degli Studi Federico II, Via Pansini, 5, Napoli
  - Istituto di Scienze Neurologiche Università di Catania, Via Santa Sofia, 78, Catania
  - Ospedale Bellaria Maggiore, Via Toscana Nazionale, 17/19, Bologna
  - Azienda Ospedaliera Careggi - Università degli Studi, Viale Giovan Battista Morgagni, 85, Firenze
- Portugal (5):
  - Hospital Fernando Fonseca, Amadora
  - Hospitais da Universidade de Coimbra, Av. Dr. Bissaya Barreto, Coimbra
  - Hospital Sto. António dos, Capuchos
  - Hospital de São João, Porto
  - Hospital de S. Bernardo, Rua Camilo Castelo Branco, Setubal
- South Korea (4):
  - National Cancer Center, 809 Madu 1-dong, Ilsan-gu, Kyunggi, Goyang
  - Samsung Medical Center, Seoul, Korea
  - Yonsei Univ. Med. Center,Severance Hospital, 134 Shinchon-dong, Suedaemoon-ku, Seoul
  - Kyung Pook National University Hospital, Taegu
- Spain (8):
  - Complejo Hospitalario Carlos Haya, Avda. Carlos Haya, S/n, Málaga
  - Hospital Universitario Virgen Macarena, Avenida Dr. Fedriani, 3, Sevilla
  - Ciutat Sanitaria I, Universitaria De Bellvitge, c/o Feixa Llarga, Hospitalet de Llobregat, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Clinico San Carlos, C/ Dr. Martin Lagos, S/n, Madrid
  - Unitat de Neuroimmunologia Clinica, Hospital Vall d'Hebron, EUI-planta 2, Pg. Vall d'Hebron 119-29, Barcelona
  - Puerta de Huerro Univeristy Hospital, San Martin de Porres, 4, Madrid
  - Hospital Universitario La Fe., Valencia
- Switzerland (2):
  - Universitätsspital Zuerich, Neurologische Klinik, Frauenklinikstrasse 26, Zuerich
  - Universitätsspital Basel, Neurochirugishen Poliklinik, Petersgraben 4, Basel
- United Kingdom (4):
  - Novartis, Investigational Site
  - Charing Cross Hospital, London
  - The Walton Centre for Neurology and Neurosurgery, Lower Lane, Fazakerly, Liverpool
  - Norfolk & Norwich University Hospital, Norwick

REFERENCES:
- [Derived] Cohen JA, Khatri B, Barkhof F, Comi G, Hartung HP, Montalban X, Pelletier J, Stites T, Ritter S, von Rosenstiel P, Tomic D, Kappos L; TRANSFORMS (TRial Assessing injectable interferoN vS. FTY720 Oral in RRMS) Study Group. Long-term (up to 4.5 years) treatment with fingolimod in multiple sclerosis: results from the extension of the randomised TRANSFORMS study. J Neurol Neurosurg Psychiatry. 2016 May;87(5):468-75. doi: 10.1136/jnnp-2015-310597. Epub 2015 Jun 25. PMID 26111826
- [Derived] Khatri BO, Pelletier J, Kappos L, Hartung HP, Comi G, Barkhof F, von Rosenstiel P, Meng X, Grinspan A, Hashmonay R, Cohen JA; TRANSFORMS Study Group. Effect of prior treatment status and reasons for discontinuation on the efficacy and safety of fingolimod vs. interferon beta-1a intramuscular: Subgroup analyses of the Trial Assessing Injectable Interferon vs. Fingolimod Oral in Relapsing-Remitting Multiple Sclerosis (TRANSFORMS). Mult Scler Relat Disord. 2014 May;3(3):355-63. doi: 10.1016/j.msard.2013.11.006. Epub 2013 Dec 12. PMID 25876473
- [Derived] Chinea Martinez AR, Correale J, Coyle PK, Meng X, Tenenbaum N. Efficacy and safety of fingolimod in Hispanic patients with multiple sclerosis: pooled clinical trial analyses. Adv Ther. 2014 Oct;31(10):1072-81. doi: 10.1007/s12325-014-0154-4. Epub 2014 Sep 23. PMID 25245812
- [Derived] Zarbin MA, Jampol LM, Jager RD, Reder AT, Francis G, Collins W, Tang D, Zhang X. Ophthalmic evaluations in clinical studies of fingolimod (FTY720) in multiple sclerosis. Ophthalmology. 2013 Jul;120(7):1432-9. doi: 10.1016/j.ophtha.2012.12.040. Epub 2013 Mar 24. PMID 23531349
- [Derived] Khatri B, Barkhof F, Comi G, Hartung HP, Kappos L, Montalban X, Pelletier J, Stites T, Wu S, Holdbrook F, Zhang-Auberson L, Francis G, Cohen JA; TRANSFORMS Study Group. Comparison of fingolimod with interferon beta-1a in relapsing-remitting multiple sclerosis: a randomised extension of the TRANSFORMS study. Lancet Neurol. 2011 Jun;10(6):520-9. doi: 10.1016/S1474-4422(11)70099-0. Epub 2011 May 13. PMID 21571593
- [Derived] Twiss J, Doward LC, McKenna SP, Eckert B. Interpreting scores on multiple sclerosis-specific patient reported outcome measures (the PRIMUS and U-FIS). Health Qual Life Outcomes. 2010 Oct 11;8:117. doi: 10.1186/1477-7525-8-117. PMID 20937112
- [Derived] Cohen JA, Barkhof F, Comi G, Hartung HP, Khatri BO, Montalban X, Pelletier J, Capra R, Gallo P, Izquierdo G, Tiel-Wilck K, de Vera A, Jin J, Stites T, Wu S, Aradhye S, Kappos L; TRANSFORMS Study Group. Oral fingolimod or intramuscular interferon for relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):402-15. doi: 10.1056/NEJMoa0907839. Epub 2010 Jan 20. PMID 20089954
- See also: Fingolimod clinical trials information website — http://www.msclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients randomized in the Core Phase (CP) to receive 0.5 mg or 1.25 mg fingolimod received the same dose in the Extension Phase (EP). Patients randomized to receive interferon-β-1a in the CP were re-randomized to receive either 0.5 mg or 1.25 mg fingolimod in a 1:1 ratio in the EP. Upon protocol amendment, all patients received 0.5 mg fingolimod.
Groups:
- Fingolimod 1.25 mg: Patients self-administered fingolimod 1.25 mg capsules orally once daily. In addition, they self-administered an interferon β-1a placebo intramuscular (im) injection once weekly.
- Fingolimod 0.5 mg: Patients self-administered fingolimod 0.5 mg capsules orally once daily. In addition, they self-administered an interferon β-1a placebo intramuscular (im) injection once weekly.
- Interferon β-1a 30 µg: Patients self-administered interferon β-1a 30 μg in an intramuscular (im) injection once weekly. In addition, they self-administered a fingolimod placebo capsule orally once daily.
- Interferon β-1a/Fingolimod 1.25 mg: Patients who received Interferon β-1a 30 µg in the core phase of the study were randomized to receive self-administered fingolimod 1.25 mg capsules orally once daily.
- Interferon β-1a/Fingolimod 0.5 mg: Patients who received Interferon β-1a 30 µg in the core phase of the study were randomized to receive self-administered fingolimod 0.5 mg capsules orally once daily.
Period: Core Phase of Study
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a 30 µg | Interferon β-1a/Fingolimod 1.25 mg | Interferon β-1a/Fingolimod 0.5 mg
Started | 426 | 431 | 435 | 0 (This group was formed at the beginning of the extension phase of the study.) | 0 (This group was formed at the beginning of the extension phase of the study.)
Completed | 369 (On study drug: 358, Off study drug: 11) | 398 (On study drug: 385, Off study drug: 13) | 386 (On study drug: 380, Off study drug: 6) | 0 | 0
Not Completed | 57 | 33 | 49 | 0 | 0
Not completed — Adverse Event | 26 | 9 | 9 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 9 | 16 | 0 | 0
Not completed — Administrative Problems | 6 | 2 | 7 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 7 | 0 | 0
Not completed — Abnormal laboratory value(s) | 4 | 6 | 1 | 0 | 0
Not completed — Abnormal test procedure result(s) | 4 | 3 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 4 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0
Period: Extension Phase of Study
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a 30 µg | Interferon β-1a/Fingolimod 1.25 mg | Interferon β-1a/Fingolimod 0.5 mg
Started | 330 (Entry into the extension phase of the study was optional.) | 357 (Entry into the extension phase of the study was optional.) | 0 (This group did not exist in the extension phase of the study.) | 176 (Entry into the extension phase of the study was optional.) | 167 (Entry into the extension phase of the study was optional.)
Received Study Drug | 330 | 356 | 0 | 174 | 167
Completed | 245 | 281 | 0 | 123 | 123
Not Completed | 85 | 76 | 0 | 53 | 44
Not completed — Subject did not receive study drug | 0 | 1 | 0 | 2 | 0
Not completed — Subject withdrew consent | 26 | 31 | 0 | 12 | 15
Not completed — Adverse Event | 21 | 22 | 0 | 19 | 7
Not completed — Abnormal laboratory value(s) | 14 | 13 | 0 | 13 | 4
Not completed — Unsatisfactory therapeutic effect | 13 | 7 | 0 | 4 | 9
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 3
Not completed — Subject no longer requires study drug | 4 | 0 | 0 | 0 | 2
Not completed — Administrative problems | 3 | 0 | 0 | 1 | 1
Not completed — Abnormal test procedure result(s) | 0 | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a 30 µg | Interferon β-1a/Fingolimod 1.25 mg | Interferon β-1a/Fingolimod 0.5 mg | Total
Number analyzed (Participants) | 426 | 431 | 435 | 174 | 167 | 1633
Age, Continuous [Mean (Standard Deviation); unit: years] — Core phase of study. Total number of patients is 1292. Demographics are based on the randomized population.
  years | 35.8 (8.39) | 36.7 (8.81) | 36.0 (8.29) | NA (NA) — This group did not exist in the core phase of the study. | NA (NA) — This group did not exist in the core phase of the study. | 36.2 (8.50)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Extension phase of study. The number of patients in the optional extension phase was less than the overall number of baseline participants who started the study. Total number of patients is 1027. Demographics are based on the intent-to-treat population.
  Years | 35.5 (8.42) | 36.5 (8.67) | NA (NA) — This group did not exist in the extension phase of the study. | 36.1 (8.11) | 36.1 (8.59) | 36.0 (8.48)
Age, Customized [Number; unit: Participants] — Core phase of study. Total number of patients is 1292. Demographics are based on the randomized population.
  Participants
    < 18 | 0 | 0 | 0 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | 0
    18-30 | 125 | 117 | 113 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | 355
    31-40 | 160 | 150 | 185 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | 495
    41-55 | 141 | 164 | 137 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | 442
    > 55 | 0 | 0 | 0 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | 0
Age, Customized [Number; unit: Participants] — Extension phase of study. The number of patients in the optional extension phase was less than the overall number of baseline participants who started the study. Total number of patients is 1027. Demographics are based on the intent-to-treat population.
  Participants
    < 18 | 0 | 0 | NA — This group did not exist in the extension phase of the study. | 0 | 0 | 0
    18-30 | 100 | 98 | NA — This group did not exist in the extension phase of the study. | 39 | 48 | 285
    31-40 | 122 | 127 | NA — This group did not exist in the extension phase of the study. | 83 | 62 | 394
    41-55 | 108 | 131 | NA — This group did not exist in the extension phase of the study. | 52 | 57 | 348
    >55 | 0 | 0 | NA — This group did not exist in the extension phase of the study. | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Core phase of study. Total number of patients is 1292. Demographics are based on the randomized population.
  Participants
    Female | 293 | 282 | 295 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 133 | 149 | 140 | NA — This group did not exist in the core phase of the study. | NA — This group did not exist in the core phase of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: Participants] — Extension phase of study. The number of patients in the optional extension phase was less than the overall number of baseline participants who started the study. Total number of patients is 1027. Demographics are based on the intent-to-treat population.
  Participants
    Female | 227 | 235 | NA — This group did not exist in the extension phase of the study. | 114 | 109 | 685
    Male | 103 | 121 | NA — This group did not exist in the extension phase of the study. | 60 | 58 | 342

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Aggregate Relapse Rate (ARR) in the Core Phase of the Study
Description: The ARR is defined as the number of confirmed relapses in a year. A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection. The annualized ARR for each treatment group was calculated using negative binomial regression adjusted by treatment, country, number of relapses in the previous 2 years, and the baseline Expanded Disability Status Scale score.
Time Frame: Baseline to Month 12
Population: Intent-to-treat population (ITT): All patients who were randomized and received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Estimate relapses per year
Groups:
- Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg: Patients received Interferon β-1a 30 µg in the core phase of the study (Baseline to Month 12) and were then randomized to receive self administered fingolimod capsules orally once daily, either 1.25 or 0.5 mg, for the remainder of the study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 420 | 429 | 431
Estimate relapses per year | 0.203 [0.157 to 0.264] | 0.161 [0.122 to 0.212] | 0.331 [0.262 to 0.417]

2. Secondary Outcome: Number of New or Newly Enlarged T2 Lesions in Comparison With Baseline in the Core Phase of the Study
Description: The number of new or newly enlarged T2 lesions in comparison to baseline was assessed with T2-weighted magnetic resonance image (MRI) scans. A T2-weighted MRI scan utilizes particular values of the echo time (TE) and the repetition time (TR) parameters of image acquisition. Inflammation and tissue damage are seen as bright areas in T2 images and are often referred to as T2 lesions. T2-weighted MRI scans are a sensitive way to evaluate the brain for demyelinating diseases, such as multiple sclerosis.
Time Frame: Baseline to Month 12
Population: Intent-to-treat population (ITT): All randomized patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 420 | 429 | 431
T2 lesions | 1.6 (3.23) | 1.6 (3.16) | 2.6 (5.50)

3. Secondary Outcome: Percentage of Participants Free of 3-month Disability Progression Assessed With the Expanded Disability Status Scale (EDSS) at the End of the Core Phase of the Study
Description: The EDSS is a scale for assessing disability in 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, other functions). An overall score ranging from 0 (normal) to 10 (death due to MS) is calculated. Disability progression was determined by the EDSS score based on the following criteria: One point increase from baseline in patients with baseline EDSS score from 0 to 5.0; or half a point increase in patients with baseline EDSS score of 5.5 or above. Percent of patients free of disability progression was calculated using the Kaplan-Meier method.
Time Frame: Baseline to Month 12
Population: Intent-to-treat population (ITT): All randomized patients who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 420 | 429 | 431
Percentage of participants | 93.3 [90.92 to 95.77] | 94.1 [91.82 to 96.33] | 92.1 [89.45 to 94.66]

4. Secondary Outcome: Estimated Annualized Aggregate Relapse Rate (ARR) in the Core and Extension Phases of the Study
Description: as for outcome 1
Time Frame: Month 0 to end of study (up to approximately 4.5 years)
Population: Intent-to-treat population (ITT): All patients who were randomized and received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Estimated relapses per year
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 420 | 429 | 431
Estimated relapses per year
  Month 12 to Month 24, n=330, 356, 341 | 0.156 [0.114 to 0.214] | 0.182 [0.138 to 0.242] | 0.266 [0.207 to 0.341]
  Month 24 to Month 36, n=287, 321, 293 | 0.116 [0.079 to 0.169] | 0.110 [0.076 to 0.160] | 0.121 [0.084 to 0.176]
  Month 36 to Month 48, n=267, 303, 271 | NA [NA to NA] — Not estimable due to sparse data. | NA [NA to NA] — Not estimable due to sparse data. | NA [NA to NA] — Not estimable due to sparse data.
  Month 48 to end of study, n=36, 38, 29 | NA [NA to NA] — Not estimable due to sparse data. | NA [NA to NA] — Not estimable due to sparse data. | NA [NA to NA] — Not estimable due to sparse data.
  Month 0 to end of study, n=420, 429, 431 | 0.192 [0.160 to 0.229] | 0.166 [0.139 to 0.199] | 0.271 [0.230 to 0.318]

5. Secondary Outcome: Number of New or Newly Enlarged T2 Lesions in the Extension Phase of the Study
Description: as for outcome 2
Time Frame: Month 12 to end of study (up to approximately 3.5 years)
Population: Intent-to-treat population (ITT): All randomized patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 279 | 317 | 288
T2 lesions
  Month 12 to Month 24 | 1.08 (2.644) | 0.87 (1.624) | 0.97 (1.923)
  Month 24 to Month 36, n=255, 289, 258 | 1.40 (3.418) | 1.04 (4.408) | 0.72 (1.733)
  Month 36 to Month 48, n=36, 34, 35 | 0.97 (1.682) | 0.59 (1.438) | 0.49 (1.483)
  Last MRI scan to end of study, n=275, 309, 290 | 1.75 (7.248) | 0.86 (2.674) | 1.03 (4.350)

6. Secondary Outcome: Percentage of Participants Free of 3-month and 6-month Disability Progression Assessed With the Expanded Disability Status Scale (EDSS) at the End of the Extension Phase of the Study
Description: as for outcome 3
Time Frame: Baseline to end of study (up to approximately 4.5 years)
Population: Intent-to-treat population (ITT): All randomized patients who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Interferon β-1a µg/Fingolimod 1.25 or 0.5 mg
Number analyzed (Participants) | 420 | 429 | 431
Percentage of participants
  Free of 3-month progression | 67.01 [57.26 to 95.77] | 71.28 [63.69 to 78.87] | 73.40 [68.56 to 78.23]
  Free of 6-month progression | 79.54 [75.07 to 84.00] | 79.76 [75.53 to 83.98] | 81.61 [77.39 to 85.83]

ADVERSE EVENTS:
Groups:
- COR FTY720 1.25 mg: COR FTY720 1.25 mg
- COR FTY720 0.5 mg: COR FTY720 0.5 mg
- COR Interferon Beta-1a: COR Interferon beta-1a
- EXT FTY720 1.25 mg: EXT FTY720 1.25 mg
- EXT FTY720 0.5 mg: EXT FTY720 0.5 mg
Arm/Group | COR FTY720 1.25 mg | COR FTY720 0.5 mg | COR Interferon Beta-1a | EXT FTY720 1.25 mg | EXT FTY720 0.5 mg
Serious Adverse Events (participants affected / at risk) | 45/420 | 30/429 | 25/431 | 77/504 | 76/523
Other Adverse Events (participants affected / at risk) | 310/420 | 302/429 | 359/431 | 446/504 | 439/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COR FTY720 1.25 mg (N=420) | COR FTY720 0.5 mg (N=429) | COR Interferon Beta-1a (N=431) | EXT FTY720 1.25 mg (N=504) | EXT FTY720 0.5 mg (N=523)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 2 | 1 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 3 | 1 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 8 | 1 | 0 | 3 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Congenital absence of cranial vault (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 4 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular oedema (Eye disorders) | 1 | 1 | 0 | 2 | 1
Tolosa-Hunt syndrome (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abasia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 2 | 0
Complication of device insertion (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 4
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abscess sweat gland (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Administration site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0 | 2 | 1 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Encephalitis herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 4 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Papilloma viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Septic encephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Complicated fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 0
Human papilloma virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 4 | 7
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1 | 2
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Critical illness polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dural fistula (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 1 | 4 | 6
Nerve root lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Progressive relapsing multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sensorimotor disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal cord ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 2
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Infertility (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COR FTY720 1.25 mg (N=420) | COR FTY720 0.5 mg (N=429) | COR Interferon Beta-1a (N=431) | EXT FTY720 1.25 mg (N=504) | EXT FTY720 0.5 mg (N=523)
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 108 | 77
Diarrhoea (Gastrointestinal disorders) | 35 | 32 | 21 | 48 | 50
Nausea (Gastrointestinal disorders) | 29 | 40 | 29 | 37 | 36
Toothache (Gastrointestinal disorders) | 18 | 12 | 9 | 13 | 33
Fatigue (General disorders) | 60 | 44 | 45 | 39 | 40
Influenza like illness (General disorders) | 15 | 15 | 158 | 24 | 18
Pyrexia (General disorders) | 14 | 18 | 76 | 33 | 30
Bronchitis (Infections and infestations) | 19 | 20 | 11 | 39 | 49
Gastroenteritis (Infections and infestations) | 12 | 10 | 11 | 31 | 36
Influenza (Infections and infestations) | 28 | 29 | 32 | 44 | 52
Nasopharyngitis (Infections and infestations) | 93 | 88 | 88 | 158 | 162
Oral herpes (Infections and infestations) | 9 | 3 | 7 | 36 | 34
Pharyngitis (Infections and infestations) | 19 | 13 | 13 | 20 | 31
Sinusitis (Infections and infestations) | 18 | 10 | 11 | 34 | 36
Upper respiratory tract infection (Infections and infestations) | 36 | 31 | 27 | 75 | 59
Urinary tract infection (Infections and infestations) | 24 | 26 | 21 | 49 | 58
Alanine aminotransferase increased (Investigations) | 24 | 28 | 8 | 44 | 34
Gamma-glutamyltransferase increased (Investigations) | 19 | 14 | 1 | 32 | 25
Lymphocyte count decreased (Investigations) | 1 | 2 | 0 | 72 | 42
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 10 | 3 | 19 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 12 | 24 | 38 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 26 | 23 | 60 | 53
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 14 | 44 | 15 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 21 | 28 | 39 | 27
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 42 | 28 | 24 | 53 | 51
Dizziness (Nervous system disorders) | 23 | 26 | 21 | 25 | 23
Headache (Nervous system disorders) | 96 | 99 | 88 | 86 | 107
Depression (Psychiatric disorders) | 18 | 21 | 32 | 40 | 44
Insomnia (Psychiatric disorders) | 19 | 17 | 13 | 32 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 20 | 16 | 54 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 8 | 7 | 17 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 17 | 15 | 31 | 38
Hypertension (Vascular disorders) | 21 | 16 | 8 | 37 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.